CLINICAL TRIAL: NCT05815862
Title: A Multi-cohort, Randomized, Open, Multicenter Phase II Study to Evaluate the Efficacy and Safety of AL2846 Capsules in Treated Subjects With Advanced Solid Tumors
Brief Title: Clinical Study of AL2846 Capsules in the Treatment of Advanced Lung Tumor and Advanced Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AL2846-II-03
Record Dates: First submitted 2023-04-04; First posted 2023-04-18 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Advanced Lung Cancer; Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AL2846 capsule (Experimental): orally administer AL2846 capsules monotherapy, 28 days as a treatment cycle.
  Interventions: Drug: AL2846 capsule

INTERVENTIONS:
Drug: AL2846 capsule — AL2846 is a multi-target tyrosine kinase inhibitor.

SUMMARY:
This is a multi-cohort, randomized, open, multicenter Phase II study to evaluate the efficacy and safety of AL2846 capsules in patients with advanced lung cancer and ovarian cancer. Objective response rate (ORR) and progression-free survival (PFS) are the primary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with advanced lung cancer or ovarian cancer confirmed by histopathology or cytology;
* Age: 18~75 years old (when signing the informed consent form); Eastern Cooperative Oncology Group (ECOG) score: 0-1;
* At least one measurable lesion according to Response Evaluation Criteria in Solid Tumours (RECIST) 1.1;
* Normal function of main organs
* The serum Human Chorionic Gonadotropin (HCG) test of female patients of childbearing age must be negative within 7 days before study enrollment and must be non-lactating; The patient should agree to use contraception during the study period and within 6 months after the end of the study period;Male subjects should agree to use contraception during the study period and for 6 months after the study period ends;
* The patient voluntarily joined the study and signed the informed consent form, with good compliance.

Exclusion Criteria:

* Combined with the following diseases or medical history:

  1. Other malignant tumors have occurred or are present at the same time within<3 years before the first administration.
  2. Inability to tolerate multiple factors affecting oral medication due to any reason;
  3. Common Terminology Criteria for Adverse Events (CTCAE) 5.0 > grade 1 therapeutic toxicity caused by any previous treatment that has not been completely relieved, excluding hair loss;
  4. Major surgical treatment or obvious traumatic injury was received within 4 weeks before the first administration;
  5. The presence of unhealed wounds, fractures, gastric and duodenal active ulcers, persistent positive fecal occult-blood, ulcerative colitis, or other conditions determined by investigators that may cause gastrointestinal bleeding or perforation;
  6. Arteriovenous thrombosis, such as cerebrovascular accident (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc., occurred within 6 months before the first medication;
  7. Those who have a history of psychotropic drug abuse and cannot abstain or have mental disorders;
  8. Subjects with any severe and/or uncontrollable disease；
* Tumor related symptoms and treatment:

  1. Had received chemotherapy, radiation, or other anticancer therapy within 4 weeks prior to first dose;
  2. Within 2 weeks before the first dose, received Chinese Traditional drugs with anti-tumor indications specified in theNational Medical Products Administration (NMPA) approved drug instructions
  3. Previously treated with anti-angiogenic drugs such as Cabozantinib, Anlotinib, Endostar and Bevacizumab;
  4. Imaging Computed Tomography (CT)or Magnetic Resonance Imaging (MRI) shows that the tumor has invaded important blood vessels or the investigator determines that the tumor is highly likely to invade important blood vessels and cause fatal massive bleeding during the follow-up study;
  5. There is a history of interstitial lung disease, severe impairment of lung function, severe pulmonary fibrosis, severe radiation pneumonia, drug-induced lung disease, and evidence of severe active lung inflammation indicated by chest CT examination during screening;
  6. There are uncontrolled pleural effusion, ascites and moderate or above pericardial effusion requiring repeated drainage;
  7. Patients with brain metastases accompanied by symptoms or symptoms controlled for less than 2 weeks;
* Patients who have participated in and used other antitumor investigational drugs within 4 weeks before the first dose;
* Central squamous cell carcinoma (lung cancer subjects) with great risk of hemoptysis;
* Patients with concomitant diseases that, in the opinion of the investigators, seriously endanger the safety of the patients or affect the completion of the study, or who are not suitable for inclusion for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Objective remission rate (ORR) | From baseline up to 12 months.
  ORR is defined as the percentage of subjects in complete remission (CR), partial remission (PR), and disease stability (SD).
Progression free survival (PFS) | From baseline up to 12 months.
  PFS is defined as the time from randomization to the first recorded progressive disease (PD) or death from any cause.

SECONDARY OUTCOMES:
Disease control rate (DCR) | From baseline up to 12 months.
  Percentage of subjects achieving complete response (CR) and partial response (PR).
Duration of remission (DOR) | From baseline up to 12 months.
  The time from the first evaluation as CR or PR to the first evaluation as PD or death from any cause.
Overall survival (OS) | From baseline to the death events, assessed up to 3 years.
  Time from the first administration to death from any cause.
Adverse events (AEs) rate | From baseline to 28 days after the last dose or initiation of a new antineoplastic therapy (whichever comes first).
  Occurrence of all adverse events, regardless of whether there was a causal relation with the studied drug.
Peak concentration (Cmax) | Pre-dose, 30 minutes, 1 hours, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 12 hours and 24 hours after dose on Day 1 and Day 28 of Cycle 1. Pre-dose on Day 7, Day 14 and 21 of cycle 1. Each cycle is 28 days.
  Maximum plasma drug concentration
Time to peak concentration (Tmax) | Pre-dose, 30 minutes, 1 hours, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 12 hours and 24 hours after dose on Day 1 and Day 28 of Cycle 1. Pre-dose on Day 7, Day 14 and 21 of cycle 1. Each cycle is 28 days.
  Time to reach peak plasma drug concentration after dose.
Clearance half life (t1/2) | Pre-dose, 30 minutes, 1 hours, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 12 hours and 24 hours after dose on Day 1 and Day 28 of Cycle 1. Pre-dose on Day 7, Day 14 and 21 of cycle 1. Each cycle is 28 days.
  The time it takes for the drug concentration in the body to drop by half
Area under blood concentration-time curve (AUC) | Pre-dose, 30 minutes, 1 hours, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 12 hours and 24 hours after dose on Day 1 and Day 28 of Cycle 1. Pre-dose on Day 7, Day 14 and 21 of cycle 1. Each cycle is 28 days.
  After administration, the area under the curve is obtained using the blood drug concentration as the ordinate and time as the abscissa.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - Shanghai Pulmonary Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No